CLINICAL TRIAL: NCT01777165
Title: A Phase 2b, Randomized, Double-Blind,Placebo-Controlled, Safety and Efficacy Trial of Multiple Dosing Regimens of ABT-719 for the Prevention of Acute Kidney Injury in Subjects Undergoing High Risk Cardiac Surgery
Brief Title: A Safety and Efficacy Trial of Multiple Dosing Regimens of ABT-719 for the Prevention of Acute Kidney Injury in Subjects Undergoing High Risk Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M13-796; 2012-003942-33 (EudraCT Number)
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Acute Kidney Injury
Keywords: GFR; Acute Kidney Injury; High Risk cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — ABT 719

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 ABT-719 lower dose (Experimental)
  Interventions: Drug: ABT-719
- Arm 2 ABT-719 intermediate dose (Experimental)
  Interventions: Drug: ABT-719
- Arm 3 ABT-719 higher dose (Experimental)
  Interventions: Drug: ABT-719
- Arm 4 placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-719 — 1 arm of ABT-719 higher dose, 1 arm of ABT-719 intermediate dose, and 1 arm ABT-719 lower dose
  Arms: Arm 1 ABT-719 lower dose; Arm 2 ABT-719 intermediate dose; Arm 3 ABT-719 higher dose
Drug: Placebo — Placebo infusion
  Arms: Arm 4 placebo

SUMMARY:
This study will evaluate the safety and efficacy of ABT-719 in preventing acute kidney injury in patients undergoing high risk cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be male or female, age greater than or equal to 18 years old.
* Subjects must have stable renal function, per Investigator discretion and no known increase in serum creatinine of greater than or equal to 0.3 mg during the preceding 4 weeks.
* Subjects with estimated glomerular filtration rate less than or equal to 60 mL/min/1.73 m2 who require intravascular iodinated contrast within 48 hours of the day of surgery, will only be included if there is no known serum creatinine increase greater than or equal to 0.3 mg.
* Subjects must be undergoing a pre-defined on-pump cardiac surgery meeting one of the following acute kidney injury risk factors:
* Subject is undergoing combined coronary artery bypass grafting (CABG) surgery and surgery of one or more cardiac valve (valve(s) surgery), or
* Subject is undergoing surgery of more than one cardiac valve (valves surgery), or
* Subject is undergoing surgery of the aortic root or ascending part of the aorta, or
* Subject is undergoing surgery of the aortic root or ascending part of the aorta, combined with coronary artery bypass graft and/or valve(s) surgery, or
* Subject has an estimated glomerular filtration rate greater than or equal to 16 mL/min/1.73 m2 and less than or equal to 59 mL/min/1.73 m2 as determined by Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) formula at Screening, and is undergoing coronary artery bypass graft or single valve surgery.

Exclusion Criteria:

* Has an eGFR less than or equal to 15 mL/min/1.73 m2.
* Cardiac surgery to be performed without cardiopulmonary bypass.
* Has ongoing sepsis or history of sepsis within the last 2 weeks or untreated diagnosed infection prior to Screening visit. Sepsis is defined as presence of a confirmed pathogen, along with fever or hypothermia, and hypoperfusion or hypotension.
* Has known or documented RIFLE "R" or AKIN "Stage I" within the previous 4 weeks.
* Recently received (within the last 10 weeks) or is anticipated to receive chemotherapy which can interfere with kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of patients developing acute kidney injury based on the Acute Kidney Injury Network (AKIN) scoring criteria by comparing the ABT-719 dose groups versus placebo group. | Up through Day 7

SECONDARY OUTCOMES:
Proportion of subjects developing at least one of the composite events: death, needing renal replacement therapy, or having greater than or equal to 25 percent reduction in estimated glomerular filtration rate or measured glomerular filtration rate | Up through Day 90
Proportion of subjects developing at least one of the composite events: death, needing renal replacement therapy, or having greater than or equal to 25 percent reduction in serum creatinine based estimated glomerular filtration rate (GFR) | Up through Day 60
Proportion of subjects developing AKI as defined by the Risk, Injury, Failure, Loss, or ESRD (RIFLE) model | Up through Day 7
Proportion of subjects developing AKI as defined by the Kidney Disease Improving Global Outcomes (KDIGO) model | Up through Day 7
Changes from baseline (defined as within 24 hours of day 0) in serum creatinine (SCr) and S-Cystatin C at all study visits from baseline to Day 90 | Up through Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Ann Eldred, MD, Study Director — AbbVie
Locations (41):
- United States (38):
  - Site Reference ID/Investigator# 83739, Danbury, Connecticut
  - Site Reference ID/Investigator# 87720, Gainesville, Florida
  - Site Reference ID/Investigator# 83746, Jacksonville, Florida
  - Site Reference ID/Investigator# 83733, Jacksonville, Florida
  - Site Reference ID/Investigator# 89178, Tampa, Florida
  - Site Reference ID/Investigator# 87693, Atlanta, Georgia
  - Site Reference ID/Investigator# 87717, Augusta, Georgia
  - Site Reference ID/Investigator# 89180, Fort Wayne, Indiana
  - Site Reference ID/Investigator# 101942, Indianapolis, Indiana
  - Site Reference ID/Investigator# 85917, Lexington, Kentucky
  - Site Reference ID/Investigator# 83732, Bethesda, Maryland
  - Site Reference ID/Investigator# 83724, Boston, Massachusetts
  - Site Reference ID/Investigator# 83745, Boston, Massachusetts
  - Site Reference ID/Investigator# 83750, Grand Blanc, Michigan
  - Site Reference ID/Investigator# 83747, Petoskey, Michigan
  - Site Reference ID/Investigator# 83744, Royal Oak, Michigan
  - Site Reference ID/Investigator# 85913, Saint Paul, Minnesota
  - Site Reference ID/Investigator# 96455, St Louis, Missouri
  - Site Reference ID/Investigator# 91253, Omaha, Nebraska
  - Site Reference ID/Investigator# 93673, Newark, New Jersey
  - Site Reference ID/Investigator# 83722, New York, New York
  - Site Reference ID/Investigator# 89176, Asheville, North Carolina
  - Site Reference ID/Investigator# 83723, Durham, North Carolina
  - Site Reference ID/Investigator# 92413, Gastonia, North Carolina
  - Site Reference ID/Investigator# 87733, Winston-Salem, North Carolina
  - Site Reference ID/Investigator# 83735, Cincinnati, Ohio
  - Site Reference ID/Investigator# 91813, Columbus, Ohio
  - Site Reference ID/Investigator# 83738, Toledo, Ohio
  - Site Reference ID/Investigator# 91693, Portland, Oregon
  - Site Reference ID/Investigator# 89182, Springfield, Oregon
  - Site Reference ID/Investigator# 83734, Pittsburgh, Pennsylvania
  - Site Reference ID/Investigator# 83730, Knoxville, Tennessee
  - Site Reference ID/Investigator# 101876, Memphis, Tennessee
  - Site Reference ID/Investigator# 90614, Charlottesville, Virginia
  - Site Reference ID/Investigator# 83725, Richmond, Virginia
  - Site Reference ID/Investigator# 87714, Tacoma, Washington
  - Site Reference ID/Investigator# 91814, Madison, Wisconsin
  - Site Reference ID/Investigator# 87739, Milwaukee, Wisconsin
- Denmark (3):
  - Site Reference ID/Investigator# 94956, Aarhus N
  - Site Reference ID/Investigator# 109295, Copenhagen O
  - Site Reference ID/Investigator# 94955, Odense C

REFERENCES:
- [Result] McCullough PA, Bennett-Guerrero E, Chawla LS, Beaver T, Mehta RL, Molitoris BA, Eldred A, Ball G, Lee HJ, Houser MT, Khan S. ABT-719 for the Prevention of Acute Kidney Injury in Patients Undergoing High-Risk Cardiac Surgery: A Randomized Phase 2b Clinical Trial. J Am Heart Assoc. 2016 Aug 20;5(8):e003549. doi: 10.1161/JAHA.116.003549. PMID 27543797